CLINICAL TRIAL: NCT05801874
Title: Gait and Posture Analysis in Hemiparetic Patients Through Optoelectronic Systems, "Smart" Tools and Clinical Evaluation
Acronym: SMART-REHAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C130
Record Dates: First submitted 2023-02-26; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Stroke Sequelae; Hemiparesis; Gait Disorders, Neurologic
MeSH Terms: conditions — Paresis; Gait Disorders, Neurologic | interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemiparetic patients: Hemiparetic patients assessed during gait and stance performance by means of different instrumental tools (smart and portable device vs 3D laboratory gait analysis) in order to evidence gait pattern; kinematics, kinetics and spatio-temporal data.
  Interventions: Diagnostic Test: Movement analysis
- Healthy age matched subjects: Healthy age matched subjects assessed during gait and stance performance by means of different instrumental tools (smart and portable device vs 3D laboratory gait analysis) in order to evidence gait pattern; kinematics, kinetics and spatio-temporal data.
  Interventions: Diagnostic Test: Movement analysis

INTERVENTIONS:
Diagnostic Test: Movement analysis — Qualitative and quantitative computerized and instrumental assessment of gait and posture.

SUMMARY:
The purpose of the study is to validate the use of smart and widespread instruments to detect kinematic, kinetic and spatio-temporal parameters in gait and postural analysis in hemiparetic and healthy individuals. Device as single Microsoft sensor Kinect v2, wearable sensorized clothing and/or smartphone-type devices will be used; it is also planned to analyze and compare such parameters with those obtained through a technique of manual palpatory analysis. Finally the obtained measures will be compared with the corresponding ones obtained with Three-dimensional instrumented gait analysis (3D-GA).

ELIGIBILITY:
Inclusion Criteria:

* patient with post-stroke chronic hemiparesis (at least 6 month post-acute event)
* ability to stand erect for 30 seconds
* ability to walk with or without aids for 10 meters

Exclusion Criteria:

* Moderate/severe cognitive impairment (MMSE < 22)
* Moderate/severe depression (Hamilton Depression Scale > 20)
* Severe spasticity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Single laboratory movement analysis with different tools and tecniques
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
GPS (Gait Profile Score index) - differences between techniques | During movement analysis
  % of agreement between 3D-GA (3 dimensional Gait Analysis - optoelectronic system) and Kinect motion analysis in the detection of kinematic data about gait collected within the GPS (Gait Profile Score Index)

SECONDARY OUTCOMES:
Gait cycle values (stance and swing duration) - differences between techniques | During movement analysis
  % of agreement between 3D-GA (3 dimensional Gait Analysis - optoelectronic system) and Kinect motion analysis in the detection of Gait cycle values (stance and swing duration)

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bigoni, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy